CLINICAL TRIAL: NCT07314242
Title: A Randomized, Double-blind, Single-dummy, Positive Drug and Placebo-controlled, Parallel Group, Multicenter, Phase 2a Study to Evaluate the Efficacy and Safety of Hemay005 in Adult Participants With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Investigate the Biomarkers of Hemay005 in Adult Participants With Moderate to Severe COPD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM005COPD2S01
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Hemay005; Roflumilast

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Single-dummy, positive drug and placebo-controlled, Parallel Group design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemay005 group (Experimental): Hemay005 tablets
  Interventions: Drug: Hemay005 tablets
- Placebo group (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo tablet
- Roflumilast group (Active Comparator): Roflumilast tablets
  Interventions: Drug: Roflumilast Oral Tablet

INTERVENTIONS:
Drug: Hemay005 tablets — Subjects take Hemay005 tablets for 12 weeks.
  Arms: Hemay005 group
Drug: Roflumilast Oral Tablet — Subjects take roflumilast tablet for 12 weeks.
  Arms: Roflumilast group
Drug: Placebo tablet — Subjects take placebo tablet for 12 weeks.
  Arms: Placebo group

SUMMARY:
A Multicenter, Randomized, Double-blind, Single-dummy, positive drug and placebo-controlled, Parallel Group, Phase 2a Study to Evaluate the Efficacy and Safety of Hemay005 in Adults with Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a phase 2a, multicenter, randomized, double-blind, single-dummy, positive drug and placebo-controlled, parallel group study to evaluate the safety and efficacy of Hemay005 in adults with moderate to severe chronic obstructive pulmonary disease (COPD). Subjects will receive Hemay005 twice daily, or placebo, or positive drug roflumilast with a maximum treatment duration of 12 weeks. The study also includes an off-treatment safety follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 40 years old at the time of signing the informed consent form, both gender;
2. Subjects with an established diagnosis of COPD (according to GOLD 2025) at least 12 months before the screening visit, with chronic bronchitis (defined as productive cough for at least 3 months in each of the prior two consecutive years) and/or with chronic productive cough at least 12 months prior to screening;
3. Confirmed diagnosis of chronic obstructive pulmonary disease at the screening visit, FEV1 (forced expiratory volume in 1 second)/FVC (forced vital capacity) ratio<70% after albuterol use, and FEV1 after albuterol use>30% predicted of normal value and equal or smalled than 70% predicted value at the screening visit;
4. Subjects on regular maintenance therapy: inhaled glucocorticoids (ICS), LAMA, or LABA, or any combination thereof. Received maintenance therapy for at least 6 months prior to screening; Maintenance therapy must not change the dosage of these drugs from 28 days before signing the informed consent form until the end of the trial (16 weeks or safety visit after early withdrawal).
5. At least one of the following effective contraceptive methods should be adopted for female patients with fertility and male patients who have not undergone vasectomy during the entire study period from the date of signing the informed consent to 3 months after the last dose. Acceptable contraceptive methods in this study include: a. abstinence; b. hormones (oral intake, patch, ring, injection, implantation) combined with male condoms. This measure must be applied at least 30 days prior to the first administration of investigational drug, otherwise another acceptable method of contraception must be used; c. intra-uterine device (IUD) combined with male condoms; d. barrier method (diaphragm, cervical cap, sponge) combined with male condoms; exceptional circumstances: a) females who have been menopausal for 5 years and more, and b) surgical sterilization (proof should be provided).
6. Subjects voluntarily participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Subjects with a prior history of asthma or concurrent diagnosis of asthma, with or without active disease, are excluded.
2. Subjects with a moderate or severe COPD exacerbation i.e. resulting in the use of systemic corticosteroids (oral/IV/IM corticosteroids) and/or antibiotics or need for hospitalisation or a lower respiratory tract infection 6 weeks prior to screening.
3. Diseases that in the opinion of the investigator may interfere with clinical assessments, such as bronchiectasis, sarcoidosis, cystic fibrosis, pulmonary hypertension, interstitial lung disease, bronchiolitis, pneumonectomy, lung cancer, congestive heart failure, diffuse bronchiolitis, silicosis, etc.
4. COPD with emphysema phenotype according to the investigator's judgment and/or medical history records (emphysema phenotype is defined as alveolar destruction leading to permanent airway obstruction, in addition to cough and sputum, subjects usually have severe symptoms of dyspnea, shortness of breath, etc.); or have alpha1-antitrypsin deficiency.
5. Patients with chronic hepatitis B virus (HBV) infection (hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb) and hepatitis B core antibody (HBcAb) should be assessed for all patients during screening: patients with positive hepatitis B surface antigen (HBsAg) will be excluded; patients with HBsAg (negative), HBsAb (negative or positive) and HBcAb (positive) should be tested for HBV-DNA, and if the HBV-DNA result is positive, patient will be excluded; if the HBV-DNA result is negative, patients can be enrolled in the study.), chronic hepatitis C virus (HCV) infection (patients with positive hepatitis C virus antibody (HCVAb) excluded) or human immunodeficiency virus (HIV) infection (patients with positive human immunodeficiency virus (HIV) antibody excluded) or Syphilis (TP) infection (excluded patients with Treponema pallidum antibody (Anti-TP) positive).
6. . The investigator judged that the patient had other conditions that were not suitable for entry into this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sputum biomarkers | Change from baseline to week 4
  Alpha-2 macroglobulin, Interleukin 1b, Leukotriene B4, Myeloperoxidase, Neutrophil elastase, Interleukin 6, Interleukin 8, etc.
Sputum cell count | Change from baseline to week 4
  Total cell count Absolute and percent of neutrophils, eosinophils, macrophages and lymphocytes differential cell count.
Blood Biomarkers | Change from baseline to week 4
  Interleukin 1b, Interleukin 33, CXC motif chemokine ligand 1, Interleukin 8, Myeloperoxidase, Interleukin 6, Monocyte chemotactic protein 1, Macrophage inflammatory protein 1b, Matrix Metalloproteinase 9, etc

SECONDARY OUTCOMES:
Sputum biomarkers | Change from baseline to week 12
  Alpha-2 macroglobulin, Interleukin 1b, Leukotriene B4, Myeloperoxidase, Neutrophil elastase, Interleukin 6, Interleukin 8, etc
Sputum cell count | Change from baseline to week 12
  Total cell count Absolute and percent of neutrophils, eosinophils, macrophages and lymphocytes differential cell count.
Blood Biomarkers | Change from baseline to week 12
  Interleukin 1b, Interleukin 33, CXC motif chemokine ligand 1, Interleukin 8, Myeloperoxidase, Interleukin 6, Monocyte chemotactic protein 1, Macrophage inflammatory protein 1b, Matrix Metalloproteinase 9, etc

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tianjin Fourth Central Hospital, Tianjin
  - China People's Armed Police Force Characteristic Medical Center, Tianjin